CLINICAL TRIAL: NCT04346511
Title: Effects of Anti-Hypertensive Acupuncture Treatment on Cerebral Blood Flow Responses to Exercise in Hypertensive Humans
Brief Title: Acupuncture Treatment on Cerebral Blood Flow
Acronym: Amp-HTN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never initiated - KSP lost interest
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11943
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Real Acupuncture(RA): In a supine position with a cardboard blocking view of their legs, patients will have six, 0.25*40mm sterilized stainless steel acupuncture needles (Dongbang Acupuncture, Inc., Seoul, South Korea) inserted into six acupoints (sites ST36, LV3, KI2, bilaterally) on their lower legs. After insertion, the needles will be stimulated at 2-4Hz, 10s at each point (1min total), immediately after insertion, 5min, 10min, 15min and just before removal. After which the needles will be removed.
  Placebo (PL): Specially designed Sham acupuncture needles that are not actually penetrate the skin and activate the acupoint will be used in an identical procedure to RA. The patient would be able to feel light pressure at the site.
Who Masked: Participant
Masking Description: This study is a single-blind crossover design. Participants will be blinded in two trials. Practitioners and operators will not be allowed to communicate with the participants concerning the type of acupuncture devices. Outcome assessors and statisticians may not be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): In a supine position with a cardboard blocking view of their legs, patients will have six, 0.25*40mm sterilized stainless steel acupuncture needles (Dongbang Acupuncture, Inc., Seoul, South Korea) inserted into six acupoints (sites ST36, LV3, KI2, bilaterally) on their lower legs. After insertion, the needles will be stimulated at 2-4Hz, 10s at each point (1min total), immediately after insertion, 5min, 10min, 15min and just before removal. After which the needles will be removed.
  Interventions: Other: Acupuncture
- Sham Acupuncture (Sham Comparator): Specially designed Sham acupuncture needles that are not actually penetrate the skin and activate the acupoint will be used in an identical procedure to RA. The patient would be able to feel light pressure at the site.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Patients will have six, 0.25*40mm sterilized stainless steel acupuncture needles (Dongbang Acupuncture, Inc., Seoul, South Korea) inserted into six acupoints (sites ST36, LV3, KI2, bilaterally) on their lower legs. After insertion, the needles will be stimulated at 2-4Hz, 10s at each point (1min total), immediately after insertion, 5min, 10min, 15min and just before removal.
  Other Names: Sham Acupuncture

SUMMARY:
Cerebrovascular diseases (CVD) and neurodegenerative diseases (NDD) are both leading causes of death in the United States. Epidemiological data have shown that increased prevalence of hypertension is related to these outcomes. However, despite the strong association of poor brain health outcomes in patients with hypertension (HTN), the understanding of cerebral blood flow (CBF) regulation and treatment options for HTN remain limited. Acupuncture treatment (AT), which is considered a promising complementary and integrative modality, has been known to reduce blood pressure and improve endothelial function in HTN. However, very few studies have investigated AT's effect on cerebrovascular function and the possible neuroprotective properties directly via regulating HTN. Exercise is used as a stimulus that increases the brain's metabolism and requires cerebrovascular responses (vasodilation) to meet the new metabolism.

Therefore, the specific aim of this study is to test the hypothesis that an antihypertensive acupuncture treatment can acutely improve cerebrovascular responses in hypertensive humans during moderate exercise.

DETAILED DESCRIPTION:
After IRB approval, experiments will take place in the Human Circulation Research Laboratory in the Department of Health and Exercise on the OU Norman campus. All subjects will complete a total of 3 visits. The first is a screening visit to provide informed consent and to ensure the potential participant meets all inclusion criteria and no exclusion criteria. Once enrolled, participants will complete two experimental trials (Placebo (PL, Sham Acupuncture) or Real Acupuncture (RA), randomized) in a single-blinded crossover design. PL or RA treatment will precede testing by ~25min before to maximize acute responses. Test begins with 5 min of quiet rest where baseline measurements are taken, followed by 5 min of exercise. After exercise, subjects will be given 5 min of quiet rest.

Visit 1 (Screening day): ~1.5 hours. The screening visit will include informed consent, health history, physical activity questionnaires and blood sample. If qualified, the subject will be enrolled in the study and they will complete a maximal oxygen uptake (VO2max) cycle ergometer test to determine fitness.

Visit 2 & 3 (Study day): ~1.5 hours. Instrumentation: Subjects will be equipped with ECG for heart rate (HR), photoplethysmography for blood pressure, pulse oximeter, mouthpiece for end-tidal CO2 (PETCO2) and oxygen uptake (VO2), near-infrared spectroscopy (NIRS) for active muscle oxygenation and Transcranial Doppler (TCD) for CBF. Real Acupuncture (RA): Subjects will receive ~20 minutes of RA treatment prior to exercise. Placebo (PL): Specially designed Sham Acupuncture needles will be used in the same acupoints, for the same duration as RA.

All subjects will complete a total of 3 visits separated by a minimum of 48 hours. Each study visit will take ~1.5 hours. The investigators anticipate ~ 6 hours or less of total involvement of the participants' time.

This study is a single-blind crossover design. Participants will be blinded in two trials. Practitioners and operators will not be allowed to communicate with the participants concerning the type of acupuncture devices. Outcome assessors and statisticians may not be blinded to treatment allocation.

The key dependent variable of interest is change (delta) in cerebrovascular conductance index (CVCi = CBF/blood pressure) from rest to exercise (delta CVCi = CVCiExercise - CVCiRest). Delta CVCi is the most common assessment of vasodilation in humans as it normalizes differences in blood flow to differences in blood pressure. CVCi calculates how much blood flow is observed for a given pressure. A change in CVCi (delta CVCi) has a predictable relationship where + delta CVCi indicates vasodilation (more flow for a given pressure) and - delta CVCi indicates vasoconstriction (less flow for a given pressure). Data will be analyzed using a general linear model approach (similar to ANOVA). Based on pilot data, a total sample size of 40 (20 CON and 20 HTN) will provide a power of 0.9. A minimum of 60 participants will be to recruited to ensure statistical power is achieved.

ELIGIBILITY:
Inclusion Criteria:

Subjects will include healthy controls (CON) and Hypertension (HTN) patients between 18-65 years of age. Female participants if premenopausal will be studied in the early follicular phase of their cycle to minimize vascular effects of circulating hormones.

HTN:

1) Stage 1 hypertensive, Systolic BP (SBP) ≥ 130 mmHg and/or Diastolic BP (DBP) > 80 mmHg, and/or diagnosis of HTN, with BMI and physical activity levels ≈ CON

1. If they are on anti-hypertensive medication, the dose, type, and frequency of use will be recorded.
2. HTN with an SBP > 139 mmHg must have a medical doctor's permission to participate

CON: will be age, BMI, menstrual status for females, and physical activity matched to HTN. They must be:

1. Normotensive
2. Free of cardiovascular comorbidities.

Exclusion Criteria:

1. Diabetes
2. Coronary artery disease
3. Stroke
4. Heart attack
5. Sleep apnea
6. Tobacco use
7. Asthma
8. Pregnancy
9. Currently receiving antihypertensive acupuncture treatment
10. conditions where acupuncture might not be safe, such as metal allergy or needle-phobia. If a subject experiences severe acupuncture-associated response, it will be subject to early termination of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular Conductance Index | 5 min of moderate exercise
  Middle Cerebral Artery Blood Velocity relative to Mean Arterial Pressure (MCABV/MAP)
Middle cerebral artery blood velocity | 5 min of moderate exercise
  Velocity of blood through the middle cerebral arteries
Mean Arterial Pressure | 5 min of moderate exercise
  Integral of blood pressure waveform

SECONDARY OUTCOMES:
Heart Rate Variability | before and after acupuncture
  measure of the variation in time between each heartbeat
End-tidal CO2 | 5 min of moderate exercise
  Partial pressure carbon dioxide (CO2) at the end of an exhaled breath
Oxygen Uptake | 5 min of moderate exercise
  Volume of oxygen consumed by the body per minute
peripheral capillary oxygen saturation | 5 min of moderate exercise
  estimate of the amount of oxygen in the blood
Tissue saturation index | 5 min of moderate exercise
  estimate of the amount of oxygen in muscle
blood glucose levels | prior to enrollment
  venous blood content
blood triglyceride levels | prior to enrollment
  venous blood content
blood high density lipoprotein levels | prior to enrollment
  venous blood content
blood low density lipoprotein levels | prior to enrolment
  venous blood content

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Kellawan, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Department of Health and Exercise Science, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.